CLINICAL TRIAL: NCT02870933
Title: The Effect of Transepicardial Augmentation on Transseptal Autologous CD 133+ Bone Marrow Cell Implantation to Myocardial Perfusion in Patient Following Coronary Artery Bypass Grafting
Brief Title: Transepicardial With Transseptal Autologous CD 133+ Bone Marrow Cell Implantation in Patient Following CABG Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Tri Wisesa Soetisna, MD, MHA, Director of Human Capital and General Affairs of National Cardiac Center, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LB.02.01/VII/086/KEP.007.EV
Record Dates: First submitted 2016-08-07; First posted 2016-08-17 (Estimated); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease
Keywords: CD 133+; Transepicardial with Transseptal Implantation; CABG
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- subject (Experimental): this arm will receive Transepicardial with Transseptal CD 133+ Implantation
  Interventions: Biological: Transepicardial with Transseptal CD 133+ Implantation
- control (No Intervention): this arm will not receive Transepicardial with Transseptal CD 133+ Implantation

INTERVENTIONS:
Biological: Transepicardial with Transseptal CD 133+ Implantation — Transepicardial with Transseptal CD 133+ Implantation
  Arms: subject

SUMMARY:
Heart Failure has several etiologies and one of them is coronary artery disease. Coronary artery bypass grafting (CABG) is one of revascularizations method which has been used for decades in coronary artery disease theraphy. However, data about coronary artery bypass grafting shows that post-CABG patients still have low ejection fraction. For the last decade, there have been a lot of studies about the using of stem cells to increase heart contractility and reverse the heart remodelling process. In this study, we use CD 133+ bone marrow stem cells which has been proved to have higher angiogenesis potential. The stem cells is given during CABG by injection transepicardial and transseptal. The purpose of this study is to determine whether transpicardial and transseptal injection of CD 133+ bone marrow stem cells can improve myocardial perfusion in patient with low ejection fraction following CABG surgery.

DETAILED DESCRIPTION:
Study sample : patient with low ejection fraction indicated for CABG surgery in NCCHK who fulfill inclusion and exclusion criteria

Sampling method : first we use consecutive method to find subject with male sex and age 40-70. After that, we use simple random sampling to allocate each subject to each group.

Total samples is 13 for each group. To anticipated drop out rate 10%, total sample is 15 for each group.

Intervention and measurement :

Control group will only receive CABG surgery. Study group will receive CBAG surgery and stem cell implantation. Stem cell aspiration will be performed 1 day before CABG procedure. Before aspiration, patients will be given local anesthetic and light sedation. Stem cell will be collected from posterior iliac crest. Total aspirate 190 cc. Stem cell CD133+ will be separated using CliniMACS® Magnetic Separation Device after labelled with Magnetic microbeads - anti CD133 labelling.

Myocardial perfusion reserve index will be measure using MRI. MPRI value will be obtained globally and segmentally in each 16 ventricle segments VEGF plasma level will be measured using sandwich Enzyme-linked Immunosorbent Assay method.

Ejection fraction, left ventricle dimension, and scar size will be measured using MRI.

Quality of life will be measured using Minnesota Living With Heart Failure Questionnaire.

Statistical analysis is done using IBM SPSS Statistics version 21.0 (SPSS inc, Chicago, IL, USA). Numerical data will be presented in either mean/standard deviation or median/min-max depend on distribution of data. Hypothesis test for numeric variable is done using paired/non-paired T test or Mann-Whitney/Wilcoxon depend on normality of data. Normality test is done using Shapiro-Wilk test. Hypothesis test for category varible is done using chi-square or fischer test.

ELIGIBILITY:
Inclusion Criteria:

* patients with coronary artery disease 3 vessels disease indicated for CABG
* LVEF < 35% which has been confirmed by MRI
* Patients with akinetic or hypokineic segment, and left ventricle myocardial hypoperfusion confirmed in MRI
* has signed informed consent

Exclusion Criteria:

Emergency CABG Ungraftable coronary artery Acute myocardial Infarct (<14 days) Valve disease which need surgery repair Contraindicated for MRI High degree ventricular arrhytmia Coagulation disorder HIV positive patient, Hepatitis B + patients, HCV + patients AST/ALT > 1,5 upper normal value Creatinine > 2 g/dl. Malignancy

Drop out criteria :

Aortic cross clamp >120 minutes and CABG total time >180

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2018-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tri Wisesa Soetisna, MD, MHA, Principal Investigator — National Cardiovascular Center Harapan Kita
Locations (1):
- National Cardiovascular Center Harapan Kita, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- CABG + Transepicardial With Transseptal CD 133+ Implantation: this arm will receive CABG + Transepicardial with Transseptal CD 133+ Implantation
- Control: this arm will receive CABG only
Period: Overall Study
Arm/Group | CABG + Transepicardial With Transseptal CD 133+ Implantation | Control
Started | 15 | 15
Completed | 13 | 13
Not Completed | 2 | 2
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- CABG + Transepicardial With Transseptal CD 133+ Implantation: this arm will receive Transepicardial with Transseptal CD 133+ Implantation
- Total: Total of all reporting groups
Arm/Group | CABG + Transepicardial With Transseptal CD 133+ Implantation | Control | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.92 (8.95) | 57.46 (6.33) | 56.69 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 12 | 12 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Indonesia | 13 | 13 | 26
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Systolic blood pressure is created when the heart beats, squeezes and push blood through arteries. The unit of measure is mmHg.
  Normal range for systolic pressure is < 120 mmHg
  mmHg | 121.92 (14.37) | 126.5 (19.60) | 123.38 (17.51)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Pressure blood exerts within arteries between heart beats. Normal range for diastolic pressure is < 80 mmHg
  mmHg | 78.00 (12.03) | 72.46 (15.36) | 75.04 (13.52)
Smoking [Count of Participants; unit: Participants] — Smoking as one of coronary artery disease risk factor.
  Participants | 11 | 9 | 20
Dyslipidemia [Count of Participants; unit: Participants] — Dyslipidemia as one of coronary artery disease risk factor.
  Participants | 6 | 11 | 17
Hypertension [Count of Participants; unit: Participants] — Hypertension as one of coronary artery disease risk factor.
  Participants | 9 | 7 | 16
Menopause [Count of Participants; unit: Participants] — Menopause as one of coronary artery disease risk factor.
  Participants | 1 | 1 | 2
Diabetes [Count of Participants; unit: Participants] — Diabetes as one of coronary artery disease risk factor.
  Participants | 5 | 9 | 14
Random blood sugar level [Mean (Standard Deviation); unit: mg/dl] — The reference values for a "normal" random glucose test in an average adult are 80-140 mg/dl, between 140-2000 mg/dl is considered pre-diabetis, and >200 mg/dl is considered diabetes according ADA guidelines.
  mg/dl | 126.85 (38.89) | 136.85 (39.0) | 131.85 (38.50)
NYHA grade III-IV [Count of Participants; unit: Participants] — NYHA (New York Heart Association) is classification for heart failure. Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Participants | 3 | 4 | 7
CCS grade III-IV [Count of Participants; unit: Participants] — Canadian Cardiovascular Society grading of angina pectoris. I : Ordinary physical activity does not cause angina II: Slight limitation of ordinary activity III: Marked limitation of ordinary physical activity IV: Inability to carry on any physical activity without discomfort, anginal syndrome may be present at rest
  Participants | 1 | 2 | 3
Six minutes walk test [Mean (Standard Deviation); unit: meters] — 6-min walk test is sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
  meters | 297.08 (72.56) | 308.92 (79.37) | 303.0 (74.75)
Left Ventricle Ejection Fraction [Mean (Standard Deviation); unit: Percentage of Ejection Fraction] — Left ventricular ejection fraction (LVEF) measured by MRI. Normal range of LVEF ranges from 50% to 70%. Borderline LVEF ranges from 41% to 49% Reduced LVEF ranges < 41%
  Percentage of Ejection Fraction | 25.88 (5.66) | 30.18 (3.85) | 28.03 (5.23)
Left Ventricle End-Systolic Volume [Mean (Standard Deviation); unit: mililiters] — Left ventricle end-systolic volume is the volume of blood in a left ventricle at the end of contraction, or systole, and the beginning of filling, or diastole.
  Normal LVESV ranges is 37 - 57 mililiters.
  mililiters | 115.87 (35.94) | 141.05 (27.77) | 128.46 (33.99)
Left Ventricle End-Diastolic Volume [Mean (Standard Deviation); unit: mililiters] — Left ventricle end-diastolic volume is the volume of blood in the left ventricle at end load or filling in (diastole) or the amount of blood in the ventricle just before systole.
  Normal ranges of LVEDV is 121 - 163 mililiters
  mililiters | 156.10 (47.46) | 200.89 (37.10) | 178.5 (47.58)
Myocardial Scar Size [Mean (Standard Deviation); unit: Percentage of Scar Area] — Percentage of myocardial scar size proportion measured by MRI to quantify and define the extent/transmurality of scar tissue, the following definitions were used
  1. spatial (circumferential) extent, the number of affected segments
  2. nontransmurality, the number of segmments with a segmental scar score of 1 or 2, and transmurality, the number of segments with a segmental scar score of 3 or 4
  3. total score, summed segmental scar scores per patient divided by 17 (which reflects the damage per patient)
  Percentage of Scar Area | 27.76 (15.76) | 24.45 (13.73) | 26.11 (14.58)
Myocardial perfusion defect [Mean (Standard Deviation); unit: Percentage of Myocardial Perfusion] — Number of heart wall segments with perfusion defect measured by MRI.
  Percentage of Myocardial Perfusion | 15.76 (4.38) | 15.38 (4.87) | 15.57 (4.62)
Wall motion score index [Mean (Standard Deviation); unit: units on a scale] — Cardiac wall motion abnormality will be measured using Wall Motion Score Index with MRI. Each myocardial segment is assigned a score from 1 to 4. The 16 segment model of myocardial segmentation is recommended.
  A WMSI of 1.0 is considered normokinetic. A WMSI of 1.5 is considered mild hypokinesia A WMSI of 2.0 is considered hypokinesia A WMSI of 2.5 is considered severe hypokinesia A WMSI of 3.0 is considered akinetic.
  units on a scale | 2.32 (0.17) | 2.07 (0.31) | 2.2 (0.28)
Minnesotta Living with Heart Failure Score [Mean (Standard Deviation); unit: units on a scale] — Quality of life assessed using Minnesota Living With Heart Failure Questionnaire consist of 21 questions, to see the changes before and after intervention.
  Minimum score = 0, Maximum score = 105 Higher values represent a worse outcome
  units on a scale | 30.3 (13.73) | 21.46 (8.76) | 25.88 (12.16)
Vascular Endothelial Growth Factor [Mean (Standard Deviation); unit: pg/mL] — Cytokine that has important role for angiogenesis. Normal range for plasma VEGF is 0-115 pg/ml
  pg/mL | 46.86 (141.20) | 40.46 (40.08) | 43.66 (101.75)

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Defect Perfusion
Description: Number of heart wall segments with perfusion defect measured by MRI.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: Percentage of Myocardial Perfusion
Groups:
- Transepicardial With Transseptal CD 133+ Implantation: this arm will receive CABG + Transepicardial with Transseptal CD 133+ Implantation
Arm/Group | Transepicardial With Transseptal CD 133+ Implantation | Control
Number analyzed (Participants) | 13 | 13
Percentage of Myocardial Perfusion
  Pre-op | 15.76 (4.38) | 15.38 (4.87)
  Post-op | 2.08 (2.13) | 3.85 (5.20)

2. Primary Outcome: Left Ventricular Ejection Fraction
Description: Left ventricular ejection fraction (LVEF) measured by MRI. Normal range of LVEF ranges from 50% to 70%. Borderline LVEF ranges from 41% to 49% Reduced LVEF ranges < 41%
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Transepicardial With Transseptal CD 133+ Implantation | Control
Number analyzed (Participants) | 13 | 13
percentage of ejection fraction
  Pre-op | 25.88 (5.66) | 30.18 (3.85)
  Post-op | 34.58 (11.32) | 31.62 (7.89)

3. Secondary Outcome: Six Minutes Walking Test
Description: Quality of life will be assessed using Six minutes walking test, to see the changes of six minutes walking test before and after intervention Distances reported for healthy individuals ages 40 yo 85 years range from 400 to 700 m..
Time Frame: Baseline, 6 months
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Transepicardial With Transseptal CD 133+ Implantation | Control
Number analyzed (Participants) | 13 | 13
meters
  Pre-op | 299 [260.50 to 350.00] | 298 [255 to 371]
  Post-op | 420 [381 to 441] | 378 [335 to 414.5]

4. Secondary Outcome: Wall Motion Score Index
Description: Cardiac wall motion abnormality will be measured using Wall Motion Score Index with MRI. Each myocardial segment is assigned a score from 1 to 4. The 16 segment model of myocardial segmentation is recommended.
  A WMSI of 1.0 is considered normokinetic. A WMSI of 1.5 is considered mild hypokinesia A WMSI of 2.0 is considered hypokinesia A WMSI of 2.5 is considered severe hypokinesia A WMSI of 3.0 is considered akinetic.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transepicardial With Transseptal CD 133+ Implantation | Control
Number analyzed (Participants) | 13 | 13
score on a scale
  Pre-op | 2.32 (0.17) | 2.07 (0.31)
  Post-op | 1.82 (0.43) | 2.08 (0.28)

5. Secondary Outcome: Myocardial Scar Size
Description: Percentage of myocardial scar size proportion measured by MRI to quantify and define the extent/transmurality of scar tissue, the following definitions were used
  1. spatial (circumferential) extent, the number of affected segments
  2. nontransmurality, the number of segmments with a segmental scar score of 1 or 2, and transmurality, the number of segments with a segmental scar score of 3 or 4
  3. total score, summed segmental scar scores per patient divided by 17 (which reflects the damage per patient)
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: Percentage of Scar Area
Groups:
- subjectTransepicardial With Transseptal CD 133+ Implantation: this arm will receive CABG + Transepicardial with Transseptal CD 133+ Implantation
Arm/Group | subjectTransepicardial With Transseptal CD 133+ Implantation | Control
Number analyzed (Participants) | 13 | 13
Percentage of Scar Area
  Pre op | 27.76 (15.76) | 24.45 (13.73)
  Post op | 25.46 (12.91) | 27.32 (12.92)

6. Secondary Outcome: Vascular Endothelial Growth Factor
Description: Cytokine that has important role for angiogenesis. Normal range for plasma VEGF is 0-115 pg/ml
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Transepicardial With Transseptal CD 133+ Implantation | Control
Number analyzed (Participants) | 13 | 13
pg/ml
  Pre-op | 46.86 (141.20) | 40.46 (40.08)
  Post-op | 61.05 (63.01) | 19.88 (33.78)

7. Secondary Outcome: Left Ventricle End Systolic Volume
Description: Left ventricle end-systolic volume is the volume of blood in a left ventricle at the end of contraction, or systole, and the beginning of filling, or diastole.
  Normal LVESV ranges is 37 - 57 mililiters.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Transepicardial With Transseptal CD 133+ Implantation | Control
Number analyzed (Participants) | 13 | 13
milliliters
  Pre-op LVESV | 115.87 (35.94) | 141.05 (7.77)
  Post-op LVESV | 126.91 (86.03) | 149.33 (44.96)

8. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire
Description: Quality of life assessed using Minnesota Living With Heart Failure Questionnaire consist of 21 questions, to see the changes before and after intervention.
  Minimum score = 0, Maximum score = 105 Higher values represent a worse outcome
Time Frame: Baseline, 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Transepicardial With Transseptal CD 133+ Implantation | Control
Number analyzed (Participants) | 13 | 13
score on a scale
  Pre-op | 27 [20 to 39.5] | 23 [15 to 26]
  Post-op | 12 [4.5 to 16] | 14 [4.5 to 15.5]

9. Secondary Outcome: Left Ventricle End Diastolic Volume
Description: Left ventricle end-diastolic volume is the volume of blood in the left ventricle at end load or filling in (diastole) or the amount of blood in the ventricle just before systole.
  Normal ranges of LVEDV is 121 - 163 mililiters
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Transepicardial With Transseptal CD 133+ Implantation | Control
Number analyzed (Participants) | 13 | 13
milliliters
  Pre-op LVEDV | 156.10 (47.46) | 200.89 (37.10)
  Post-op LVEDV | 183.68 (94.99) | 219.97 (35.64)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Subject: this arm will receive CABG + Transepicardial with Transseptal CD 133+ Implantation
Arm/Group | Subject | Control
All-Cause Mortality (participants affected / at risk) | 2/13 | 1/13
Serious Adverse Events (participants affected / at risk) | 2/13 | 1/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subject (N=13) | Control (N=13)
Sepsis (Infections and infestations) | 1 | 1
Haemodynamic instability (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT02870933/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT02870933/ICF_001.pdf